CLINICAL TRIAL: NCT01591772
Title: Structural and Functional Imaging and Cognitive Functions in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-075
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cancer
Keywords: FALLOPIAN TUBE; OVARY; PERITONEUM; Quality of Life; structural MRI; functional MRI; neuropsychological assessment; 12-075
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- diagnosed with ovarian that recieved chemo
  Interventions: Other: Neuroimaging & Neuropsychological Evaluation
- healthy controls
  Interventions: Other: Neuroimaging & Neuropsychological Evaluation

INTERVENTIONS:
Other: Neuroimaging & Neuropsychological Evaluation — Will undergo structural and functional MRI scans on a Siemens 3T Magnetom Tim Trio research scanner located at the Citigroup Biomedical Imaging Center at Weill Cornell Medical Center (WCMC), which is adjacent to the MSKCC campus. Patients do not undergo routine clinical brain MRIs as part of their assessment and treatment, and the brain MRI scans to be performed in this study are for research purposes only. The MRI scan takes approximately 60 minutes to complete, and about 15 minutes will be required for instructions prior to initiating the study. The MRI studies will be reviewed by a neuroradiologist (Dr. Karimi) to rule out gross structural CNS abnormalities; in case any abnormalities considered to require clinical follow-up are detected, the subject will be contacted and referred for follow-up with their treating physician. Patients will undergo a brief neuropsychological test battery at MSKCC or at Citigroup Biomedical Imaging Center at WCMC
  Groups: diagnosed with ovarian that recieved chemo
Other: Neuroimaging & Neuropsychological Evaluation — Will undergo structural and functional MRI scans on a Siemens 3T Magnetom Tim Trio research scanner located at the Citigroup Biomedical Imaging Center at Weill Cornell Medical Center (WCMC), which is adjacent to the MSKCC campus. Patients do not undergo routine clinical brain MRIs as part of their assessment and treatment, and the brain MRI scans to be performed in this study are for research purposes only. The MRI scan takes approximately 60 minutes to complete, and about 15 minutes will be required for instructions prior to initiating the study. The MRI studies will be reviewed by a neuroradiologist (Dr. Karimi) to rule out gross structural CNS abnormalities; in case any abnormalities considered to require clinical follow-up are detected, the subject will be contacted and referred for follow-up with their treating physician. Patients will undergo a brief neuropsychological test battery at MSKCC or at Citigroup Biomedical Imaging Center at WCMC
  Groups: healthy controls

SUMMARY:
The purpose of this study is to learn about possible changes in brain anatomy and function, and in thinking abilities, such as memory skills, in patients with ovarian cancer who receive treatment with chemotherapy. Cancer patients treated with chemotherapy may experience changes in thinking abilities, and these may interfere with quality of life. Most of the research to date has involved patients with breast cancer, and there are no studies in women with ovarian cancer looking at at treatment-related changes in brain anatomy and function.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stage I-IV ovarian, peritoneal or fallopian tube cancer
* completed first-line taxane and platinum-based chemotherapy 1-4 months prior to being enrolled in the study (can be on bevacizumab maintenance)
* in remission of their disease at the time of enrollment between 21 and 70 years of age
* fluent in English
* in the judgment of the consenting professional, have capacity to give consent

Healthy Control Inclusion Criteria:

* no diagnosis of cancer except basal cell carcinoma
* between 21 and 70 years of age
* fluent in English
* has a mini-mental state exam (MMSE) score of 26 or higher
* in the judgment of the consenting professional, have capacity to give consent

Exclusion Criteria:

* active or recurrent disease, or diagnosis of another cancer (except basal cell carcinoma) as per medical records at the time of enrollment
* exposure to chemotherapy or radiation therapy for any medical condition unrelated to ovarian cancer
* on hormonal therapy at the time of enrollment
* neurological disorder or moderate to severe head trauma (loss of consciousness > 60 min)
* neurodegenerative disorders such as Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc.
* self-reported Axis I psychiatric disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia
* unable to complete cognitive tests
* with standard contraindications to MRI examinations

Healthy Control Exclusion Criteria:

* exposure to chemotherapy or radiation therapy for any medical condition
* on hormone replacement therapy at the time of enrollment
* neurological disorder or moderate to severe head trauma (loss of consciousness > 60 min)
* neurodegenerative disorders such as Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified and recruited by physicians in the Gynecologic Medical Oncology Clinic at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-04-24 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
alterations in regional brain volume | 1 year
  will undergo structural MRI scans on a Siemens 3T Magnetom Tim Trio research scanner located at the Citigroup Biomedical Imaging Center at Weill Cornell Medical Center (WCMC), which is adjacent to the MSKCC campus. Three to five T1 weighted sagittal slices are collected to localize the anterior and posterior commissures. Functional imaging: Blood Oxygenation Level-Dependent (BOLD) contrast imaging, which reflects changes in venous deoxyhemoglobin associated with neuronal activity, will be used.
dorsolateral prefrontal cortex | 1 year
  will undergo functional MRI scans on a Siemens 3T Magnetom Tim Trio research scanner located at the Citigroup Biomedical Imaging Center at Weill Cornell Medical Center (WCMC), which is adjacent to the MSKCC campus.Three to five T1 weighted sagittal slices are collected to localize the anterior and posterior commissures. Functional imaging: Blood Oxygenation Level-Dependent (BOLD) contrast imaging, which reflects changes in venous deoxyhemoglobin associated with neuronal activity, will be used.

SECONDARY OUTCOMES:
neuropsychological functions | 1 year
  Patients will undergo a brief neuropsychological test battery at MSKCC or at Citigroup Biomedical Imaging Center at WCMC. All subjects will undergo a neuropsychological evaluation including standardized tests of attention and working memory, executive functions, and memory considering that these domains have been shown to be particularly sensitive to cancer treatment-induced cognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Correa, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/